CLINICAL TRIAL: NCT06617910
Title: Treatment Outcomes and Dosimetric Analysis Comparison Between CyberKnife and VMAT Based Methods of Stereotactic Radiotherapy for Sinonasal Malignancy
Brief Title: Stereotactic Radiotherapy for Sinonasal Malignancy
Status: Active, not recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE23395C
Record Dates: First submitted 2024-09-22; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Neoplasms
Keywords: Sinonasal Malignancy; SBRT; CyberKnife
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sinonasal malignancy patients received post-operative cyberknife: Sinonasal malignancy patients in our hospital receive curative surgery. These patients received post-operative radiotheray of SBRT by cyberknife.
  Interventions: Radiation: SBRT by Cyberknife

INTERVENTIONS:
Radiation: SBRT by Cyberknife — The patients with sinonasal maliganacy receive curative surgery then receive adjuvant RT by the method of SBRT by Cyberknife.

SUMMARY:
Sinonasal Tumors are a rare type of head and neck tumor, accounting for approximately 3% of head and neck cancers. Treatment primarily involves surgical intervention, with radiation therapy as an adjunct. Due to the tumor's anatomical location near critical structures such as the eyes, optic nerves, optic chiasm, brainstem, and oral cavity, if the tumor cannot be completely resected, postoperative radiation therapy is often necessary. Given the complexity of the tumor's anatomical position, subsequent radiation therapy planning becomes more challenging, as it must balance tumor control and organ preservation. This study retrospectively analyzes patients with sinonasal tumors who received stereotactic radiosurgery (CyberKnife) at our hospital, comparing the dosimetric advantages, treatment efficacy, survival analysis, and side effects with those of volumetric modulated arc therapy (VMAT).

ELIGIBILITY:
Inclusion Criteria:

* The pathological tissue report from the endoscopic surgery at this hospital confirmed a diagnosis of malignant sinus tumor.
* Received radical stereotactic radiotherapy at this hospital.
* Pre-treatment baseline imaging (CT or MRI) was performed.
* Received radical radiotherapy at this hospital and has been under long-term follow-up with complete medical records at this hospital.

Exclusion Criteria:

* Local lymphatic metastasis and distant metastasis have been excluded by imaging examinations (cN >=1, M =1).
* Not treated with radical radiotherapy at this hospital and has been under long-term follow-up at this hospital with incomplete medical records.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sixth-generation computer-assisted radiotherapy system was introduced at this hospital in 2019. This study will attempt to analyze the dose differences between treatment plans using traditional linear accelerators and those using the computer-assisted system for patients who received stereotactic radiotherapy at this hospital over the past five years.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival, OS | Data within five years after treatment.
  Determine the start dates of surgery and radiotherapy from the hospital's medical record system, and collect data on death events, regardless of whether they are tumor-related.
Disease-Free Survival, DFS | Data within five years after treatment
  Determine the treatment start date from the hospital's medical record system, and confirm whether there is any disease recurrence or progression through follow-up data or imaging examination results.
Local Control, LC | The observation periods are 1 year, 3 years, and 5 years after treatment.
  Measure the proportion of no recurrence in the local tumor area after treatment. Researchers determine the treatment start date from the hospital's medical record system and confirm the presence or absence of local tumor recurrence through follow-up data, imaging examinations, and pathology results.
Distant Metastasis-Free Survival, DMFS | The observation periods are 1 year, 3 years,and 5 years after treatment.
  Measure the time until the occurrence of distant metastasis after treatment. Researchers first determine the treatment start date, and then assess distant metastasis through data, imaging examinations, and clinical evaluations.

SECONDARY OUTCOMES:
treatment-related side effects | complications related to treatment within 30 days
  Acute or chronic side effects caused by treatment can include radiation dermatitis, dry mouth, vision impairment, and so on.
Dosimetric Outcomes | Data for five years after treatment.
  The quality of a radiation therapy plan can be assessed through dose uniformity and dose constraints for adjacent critical organs (such as the optic nerve and brainstem). Researchers first collect dose distribution data from the treatment planning system and use dose calculation software to analyze dose uniformity indices (such as the homogeneity index) to evaluate the distribution of doses. At the same time, dose constraint standards for adjacent critical organs are established to ensure that the doses to these organs remain within safe limits during treatment. These indicators reflect the quality of the radiation therapy plan and can help researchers assess the safety and efficacy of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan